CLINICAL TRIAL: NCT04931901
Title: Paired Assessment of Two Electromyographic Neuromuscular Monitors: Stimpod NMX450X Versus Datex-Ohmeda E-NMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: StimpodVSDatex-Ohmeda
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Neuromuscular Manifestations
MeSH Terms: conditions — Neuromuscular Manifestations

STUDY DESIGN:
Intervention Model Description: Randomization per dominant and nondominant hand. So that there is an even share of number of patients with Stimpod NMX450X on dominant hand and Datex-Ohmeda E-NMT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimpod NMX450X (Experimental)
  Interventions: Device: EMG TOF device
- Datex-Ohmeda E-NMT (Active Comparator)
  Interventions: Device: EMG TOF device

INTERVENTIONS:
Device: EMG TOF device — Use of Stimpod NMX450X as an electromyographic neuromuscular monitor

SUMMARY:
After anesthesia is induced, 2 EMG TOFF devices will be placed on the patients arms, one on the right arm, the other on the left. There will be a randomization per dominant hand and nondominant hand for the placing of the devices. The devices are the Stimpod NMX450X and the Datex-Ohmeda E-NMT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old and above)
* undergoing General Anaesthesia for noncardiac surgery requiring the use of a neuromuscular blocking agent.

Exclusion Criteria:

* Use of different types of neuromuscular blocking agents for the same patient within the same surgical procedure.
* Known Neuromuscular diseases/syndromes judged to condition accurate neuromuscular monitoring.
* Known acute or chronic hepatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
TOF-ratio (percentage) | Up until 120 minutes
  TOF = Train-of-four. TOF-ratio is the ratio of the fourth muscle response to the first one. This is used to assess neuromuscular transmission. TOF% indicates fade in non-depolarizing block. We are comparing the calculated TOF ratio of the stimpod NMX to the datex-ohmeda E-NMT

SECONDARY OUTCOMES:
TOF-count (absolute number) | Up until 120 minutes.
  TOF count is the actual number of detected muscle responses. The number that is used to calculate the percentage (TOF-ratio). When the TOF count drops below 4 responses, then the TOF% cannot be calculated. We are comparing the detected muscle responses of the stimpod NMX to the datex-ohmeda E-NMT

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No